CLINICAL TRIAL: NCT04870177
Title: Phase II Study of AK112 (Anti-PD-1 and VEGF Bi-specific Antibody) in the Treatment of Advanced Gynecological Carcinoma
Brief Title: Study of AK112 in the Treatment of Advanced Gynecological Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-203
Record Dates: First submitted 2021-04-05; First posted 2021-05-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Cancer; Cancer Metastatic; Ovarian Neoplasms; Cervical Neoplasm; Endometrial Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced gynecological neoplasms (Experimental)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — AK112 infusion biweekly

SUMMARY:
A phase II study to evaluate the efficacy and safety of AK112 in subjects with advanced gynecological tumors.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent
* 18 to 75 years old of age during enrollment
* Has ECOG performance status of 0 or 1
* Has a life expectancy of at least 3 months
* Confirmed diagnosis of advanced gynaecological neoplasm
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy
* Has adequate organ functions (e.g hematology, renal, hepatic and coagulation)
* All female subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment
* Be able and willing to comply with all requirements of study participation (including all study procedures)

Exclusion Criteria:

* Known history of other malignancy (in the last 5 years) except localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, cervical carcinoma in situ, breast carcinoma in situ that has undergone curative therapy and breast carcinoma that has not recurred for > 3 years after radical surgery
* Is currently participating in a study of an investigational agent or using an investigational device 4 weeks prior to first administration of study drug
* For patients with platinum-resistant recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, prior abdominal and pelvic radiation therapy was performed
* For recurrent/metastatic endometrial carcinoma, subjects had carcinosarcomas (malignant mixed Mullerian tumors), endometrial leiomyosarcomas or other high-grade sarcomas, or endometrial stromal sarcomas
* Ovarian carcinoma of non-epithelial origin, fallopian tube cancer, primary peritoneal carcinoma (e.g., germ cell tumor); Ovarian neoplasms with low malignancy potential (e.g. borderline neoplasms)
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Previous history of immunodeficiency; HIV antibody positive; Current long-term use of systemic corticosteroids or other immunosuppressants
* Severe infection, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia, occurs within 4 weeks prior to the first administration of the study drug; Active infection with systemic anti-infective therapy (excluding antiviral therapy for hepatitis B or C) within two weeks prior to first administration of study drug
* Untreated active hepatitis B subjects; subjects with hepatitis B are required to receive anti-HBV therapy during the study period; active hepatitis C subjects
* Has undergone major surgery within 30 days prior to the first dose of study treatment
* Has known active central nervous system (CNS) metastases
* Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia. Unstable angina, myocardial infarction, congestive heart failure, or vascular disease requiring hospitalization (such as aortic aneurysm at risk of rupture), or other cardiac impairment (such as poorly controlled arrhythmias, myocardial ischemia) that may affect study drug safety evaluation within 12 months prior to first administration of study drug
* Previous history of abdominal fistula or gastrointestinal perforation associated with anti-VEGF therapy; the imaging results revealed the invasion of intestinal wall by neoplasm during screening
* During screening, imaging or clinical findings of gastrointestinal obstruction, including incomplete obstruction
* Previous history of severe bleeding or coagulation disorders; during screening, imaging showed that the neoplasm surrounded major blood vessels or had obvious necrosis and cavitation, and the investigators believed that participation in the study might increase risk of bleeding
* Has received a live virus vaccine within 30 days prior to first administration of study drug or plan to be administered during the study period
* Has known psychiatric or substance abuse disorders
* Is pregnant, breastfeeding women
* Any prior or current disease, treatment, or laboratory test abnormality that may confound the study endpoints, interfere with subjects' full participation in the study, or may not be in their best interest to participate in this study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Objective response rates (ORR) according to RECIST v1.1 in the FAS population | Up to approximately 2 years

SECONDARY OUTCOMES:
Efficacy endpoint: disease control rate (DCR) assessed according to RECIST v1.1 | Up to approximately 2 years
Efficacy endpoint: duration of response (DOR) assessed according to RECIST v1.1 | Up to approximately 2 years
Efficacy endpoint: time to response (TTR) assessed according to RECIST v1.1 | Up to approximately 2 years
Efficacy endpoint: progression-free survival (PFS) assessed according to RECIST v1.1 | Up to approximately 2 years
Efficacy endpoint: overall survival (OS) assessed according to RECIST v1.1 | Up to approximately 2 years
Serum PK concentrations of AK112 in individual subjects at different time points after AK112 administration | Up to approximately 2 years
Number of subjects with detectable anti-drug antibodies (ADA) | Up to approximately 2 years
Percentage of subjects with detectable anti-drug antibodies (ADA) | Up to approximately 2 years
Correlation between the expression of PD-L1 and the antitumor activity of AK112 in tumor tissues | Up to approximately 2 years
Correlation between microsatellite instability (MSI) and mismatch repair defect (DMMR) in tumor tissue samples from patients with endometrial cancer and the antitumor activity of AK112 | Up to approximately 2 years
The association between BRCA1/2 mutation and AK112 antitumor activity in peripheral blood samples and tumor tissues from patients with epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD, Study Chair — Qilu Hospital of Shandong University; Qi Zhou, MD, Study Chair — Chongqing University Cancer Hospital
Locations (2):
- China (2):
  - Qilu Hospital of Shandong University, Qilu, Shandong
  - Chongqing University Cancer Hospital, Chongqing